CLINICAL TRIAL: NCT07217964
Title: Evaluating Natural Matrix Protein (NMP) in Lumbar Spinal Fusion
Brief Title: Natural Matrix Protein
Acronym: NMP
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Gbolabo Sokunbi, MD, Hospital for Special Surgery, New York
Other Study IDs: 2024-2081
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-03

CONDITIONS: Degenerative Lumbar Spinal Conditions
Keywords: Lumbar; Natural Matrix Protein; Fusion; Allograft
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients (≥ 18 years old) who underwent lumbar fusion: NMP graft with interbody cage
  Interventions: Radiation: Radiographic Evaluation

INTERVENTIONS:
Radiation: Radiographic Evaluation — surgical procedure
  Other Names: Surgical

SUMMARY:
This clinical study is a non-randomized, consecutive, single-center, retrospective-prospective investigation of patients who received NMP bioimplant (Induce Biologics, Tampa, FL) in lumbar spinal fusion procedures. The purpose of this study is to assess the radiographic, clinical, and safety outcomes of Natural Matrix Protein (NMP) as a graft alternative in lumbar fusion procedures.

Utilizing the Hospital for Special Surgery's EPIC database under Institutional Review Board approval, all patients with symptomatic lumbar degenerative disc disease who failed conservative management at up to four vertebral levels between L1-S1 between February 2024 and December 2025 will be reviewed.

The inclusion criteria for the study will be adult patients (≥ 18 years old) who underwent lumbar fusion with an NMP graft and interbody cage. The exclusion criteria will include previous lumbar fusion attempts, active malignancy, concurrently under chemotherapy, active infection at time of surgery, mentally compromised, and trauma to the operated region. It is expected approximately 100 patients will fit the inclusion/exclusion criteria.

The objective of the study is to evaluate the clinical outcomes of the subjects treated with NMP

DETAILED DESCRIPTION:
Retrospective Data Collection:

Patient data was collected into a data sheet to collect specific elements that relate to safety and efficacy of the procedure utilizing this specific device system. The data elements of interest are:

Patient Summary data (where appropriate: average, sd, range):

Subject demographics Distribution of primary diagnoses

Surgical Information:

Length of constructs with note of non-contiguous constructs Levels treated Patient Assessments and Questionnaires prior to surgery Type and brand of interbody implant(s) used (if applicable) Induce and other bone graft materials used Adverse Events (defined in section 3.5) Description of adverse events Radiographic imaging at pre-operative, discharge, and follow-up time points of 6 months post-operatively (as available)

Prospective Data Collection:

Patients will be consented at their 12 month follow-up to participate in the clinical study. Clinical and radiographic data will be collected.

12 month radiographic data (SOC x-rays and CTs) Patient Assessment Questionnaires Surgeon Assessment of Patient Classification of any Secondary Surgical Procedures Adverse Events If patient has not achieved fusion, patient will be asked if they would be willing to follow-up at 24 months

Radiographic Assessment Imaging assessments will be performed by an independent imaging reviewer. The reviewer will be a musculoskeletal radiologist. The reviewer will be trained on the schedule of imaging assessments and classification systems for performing each assessment. The reviewer will not have access to clinical outcome data. Plain lateral radiographs at baseline, immediate postoperative, 6-month follow-up, 1-year follow-up, and 2-year follow-up (if available) will be utilized. All radiological measurements will be made using Sectra IDS7 (Sectra AB, Linköping, Sweden).

Fusion status on radiographs will be graded at each treated segment from an analysis of three components: bridging bone between the vertebral bodies, angular motion, and translational motion. Fusion Status measured on radiographs was derived from the qualitative assessment of bridging bone and the quantitative assessments of angular and translational Motion and in accordance to FDA guidance. The following grading system was implemented:

Not Fused: Absence of bridging bone from endplate to endplate in the intervertebral space, or angular motion > 3 degrees, or translational motion > 2 mm.

Fused: Presence of bridging bone from endplate to endplate in the intervertebral space, angular motion ≤ 3 degrees, and translational motion ≤ 2mm.

Retrospective-prospectively collected data will be recorded from subject electronic medical records

Study enrollment consists of 100 consecutive subjects who have consented to the study.

Statistical Analysis:

A performance goal methodology will be utilized to assess the primary outcome of fusion rate compared to literature controls. A literature review was conducted to find appropriate comparative studies that had similar criteria for the assessment of fusion for the performance model. The following studies are 1 level and 2 level lumbar interbody fusion studies that we used as the comparators:

Fairbank J. Re: Zigler J, Delamarter R, Spivak J, et al. Results of the prospective, randomized, multicenter Food and Drug Administration investigational device exemption study of the ProDisc-L total disc replacement versus circumferential fusion for the treatment of 1-level degenerative disc disease. Spine 2007;32:1155-62. Spine (Phila Pa 1976). 2007 Dec 1;32(25):2929-30; author reply 2930-1. doi: 10.1097/BRS.0b013e31815b84ca. PMID: 18246024.

Delamarter R, Zigler JE, Balderston RA, Cammisa FP, Goldstein JA, Spivak JM. Prospective, randomized, multicenter Food and Drug Administration investigational device exemption study of the ProDisc-L total disc replacement compared with circumferential arthrodesis for the treatment of two-level lumbar degenerative disc disease: results at twenty-four months. J Bone Joint Surg Am. 2011 Apr 20;93(8):705-15. doi: 10.2106/JBJS.I.00680. Epub 2011 Mar 11. PMID: 21398574.

Burkus JK, Heim SE, Gornet MF, Zdeblick TA. Is INFUSE bone graft superior to autograft bone? An integrated analysis of clinical trials using the LT-CAGE lumbar tapered fusion device. J Spinal Disord Tech. 2003 Apr;16(2):113-22. doi: 10.1097/00024720-200304000-00001. PMID: 12679664.

From this modelling, our primary outcome performance goal would be an 96% fusion rate with a confidence interval of 93-99%.

Sample size calculation A total sample of 101 patients is needed for this study to estimate a fusion rate of 0.96 with two-sided 95% confidence interval of (0.93,0.99).

References Fleiss, J. L., Levin, B., Paik, M.C. 2003. Statistical Methods for Rates and Proportions. Third Edition. John Wiley & Sons. New York.

Newcombe, R. G. 1998. 'Two-Sided Confidence Intervals for the Single Proportion: Comparison of Seven Methods.' Statistics in Medicine, 17, pp. 857-872.

Statistical analysis plan Counts and percentages of fusion status will be summarized. 95% confidence interval for the proportion estimate will also be calculated. VAS satisfaction and ODI score will be summarized as mean and standard deviation, or median and IQR based on the distribution of them.

ELIGIBILITY:
Inclusion Criteria:1. Patients experiencing symptomatic lumbar degenerative disc disease who failed conservative management at up to four vertebral levels between L1-S1 between February 2024 and December 2024.

2. Adult patients (≥ 18 years old) who underwent lumbar fusion with an NMP graft and interbody cage

-

Exclusion Criteria:1. Previous lumbar fusion attempts at the level of surgery (adjacent lumbar levels are acceptable) 2. Active Malignancy 3. Concurrently under chemotherapy 4. Active infection at time of surgery 5. Mentally compromised 6. Trauma to the operated region

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Radiographs | From May 2025 until May 2027
  Radiographic:
  Imaging assessments will be performed by an independent imaging reviewer. The reviewer will be a musculoskeletal radiologist trained in the schedule of imaging assessments and classification systems for performing each assessment. The reviewer will not have access to clinical outcome data. Plain lateral radiographs at baseline, immediate postoperative, 6-month follow-up, and 1-year follow-up. All radiological measurements will be made using Sectra IDS7 (Sectra AB, Linköping, Sweden).
  Fusion status on radiographs will be graded at each treated segment from an analysis of three components: bridging bone between the vertebral bodies, angular motion, and translational motion. Fusion Status measured on radiographs was derived from the qualitative assessment of bridging bone and the quantitative assessments of angular and translational Motion. The following grading system was implemented:
  Not Fused: Absence of bridging bone from endplate to endplate

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Abjornson, PhD, Study Director — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
data is aggragated for reporting

REFERENCES:
- [Background] D'Souza M, Macdonald NA, Gendreau JL, Duddleston PJ, Feng AY, Ho AL. Graft Materials and Biologics for Spinal Interbody Fusion. Biomedicines. 2019 Sep 26;7(4):75. doi: 10.3390/biomedicines7040075. PMID 31561556
- [Background] Rathbone J, Rackham M, Nielsen D, Lee SM, Hing W, Riar S, Scott-Young M. A systematic review of anterior lumbar interbody fusion (ALIF) versus posterior lumbar interbody fusion (PLIF), transforaminal lumbar interbody fusion (TLIF), posterolateral lumbar fusion (PLF). Eur Spine J. 2023 Jun;32(6):1911-1926. doi: 10.1007/s00586-023-07567-x. Epub 2023 Apr 18. PMID 37071155
- [Background] Martin BI, Mirza SK, Spina N, Spiker WR, Lawrence B, Brodke DS. Trends in Lumbar Fusion Procedure Rates and Associated Hospital Costs for Degenerative Spinal Diseases in the United States, 2004 to 2015. Spine (Phila Pa 1976). 2019 Mar 1;44(5):369-376. doi: 10.1097/BRS.0000000000002822. PMID 30074971
- [Background] Fehlings MG, Tetreault L, Nater A, Choma T, Harrop J, Mroz T, Santaguida C, Smith JS. The Aging of the Global Population: The Changing Epidemiology of Disease and Spinal Disorders. Neurosurgery. 2015 Oct;77 Suppl 4:S1-5. doi: 10.1227/NEU.0000000000000953. PMID 26378347